CLINICAL TRIAL: NCT05823272
Title: Effect of Oral Nutritional Supplement on Nutritional Status and Clinical Outcome in Gastric Cancer Patients After Total Gastrectomy
Brief Title: ONS in Gastric Cancer After Total Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Collaborators: Zhongda Hospital (Other); Shandong Provincial Hospital (Other Government); Hebei Medical University Fourth Hospital (Other); Zunyi Medical College (Other); Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Wang Xinying, Prof., Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-7-4
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
Keywords: Oral nutritional supplement; Sarcopenia; long-term nutritional status
MeSH Terms: conditions — Stomach Neoplasms; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral nutritional supplement (Experimental): In the oral nutritional supplement group, in addition to diet, and patients will also consume enteral nutrition powder (500 ml/d, 500kcal/d) lasted for 6 months after discharge.
  Interventions: Other: ONS
- control (No Intervention): In the control group, patients will receive nutrition counseling in addition to diet.

INTERVENTIONS:
Other: ONS — oral nutritional supplement
  Arms: oral nutritional supplement

SUMMARY:
Gastric cancer patients after total gastrectomy will be randomized to oral nutritional supplement group or control group at discharge. Patients will receive 6 months of oral nutritional supplement or normal diet after discharge. The primary and secondary outcomes will be collected.

DETAILED DESCRIPTION:
Gastric cancer patients after total gastrectomy at discharge, if she/he has nutrition risk (NRS2002≥3), then she/he will be randomized to oral nutritional supplement (ONS) group or control (C) group after discharge. In the ONS group, in addition to diet, and patients will also consume enteral nutritional powder (500ml/d，500kcal/d) lasted for 6 months. In the C group, patients will receive normal diet. Both groups will receive nutrition counseling.

The primary and secondary outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of patients or their legal representatives to participate in this study
2. consecutive adult (18-80 years) patients underwent radical gastrectomy (total gastrectomy)
3. nutrition Risk Screening (NRS) 2002≥3 at discharge
4. eastern Cooperative Oncology Group (ECOG) score of 0-2 at discharge
5. normal liver and kidney function

Exclusion Criteria:

1. unable to oral or consume ONS
2. allergy to any ingredient in the oral nutrition powder
3. pregnancy
4. palliative surgery or gastric stump cancer
5. congenital acquired immune deficiency disease
6. severe liver and kidney diseases including active hepatitis, cirrhosis, and uremia diabetes has developed complications or uncontrolled by medications
7. motor system diseases cannot complete grip strength measurement and 5-time chair stand test
8. have cognitive impairment, unable to complete the relevant questionnaires
9. expected to require tube feeding after discharge from the hospital

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-22 (Estimated); Primary Completion 2024-08-05 (Estimated); Study Completion 2024-08-05 (Estimated)

PRIMARY OUTCOMES:
incidence of sarcopenia 6-month after discharge | up to 6 months.
  sarcopenia is defined as low skeletal muscle mass plus low muscle strength or low physical ability.

SECONDARY OUTCOMES:
incidence of sarcopenia 1 year after discharge | up to 12 months.
  sarcopenia is defined as low skeletal muscle mass plus low muscle strength or low physical ability.
unplanned readmission rate | up to 6 months.
  readmission due to unplanned reason
toxicity of chemotherapy graded according to the CTCAE, version 5.0 | up to 6 months.
  Chemotherapy toxicity will be monitored at end of each cycle during chemotherapy by investigators, and graded according to the CTCAE, version 5.0.
Quality of life after discharge | up to 12 months.
  Quality of life assessed by EORTC QLQ-C30
Changes in BMI (weight and height will be combined to report BMI in kg/m^2) | up to 12 months.
  nutritional status after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Xinying Wang, MD, Principal Investigator — Jinling Hosptial
Locations (1):
- Jinling Hospital, China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu J, Huang C, Sun Y, Su X, Cao H, Hu J, Wang K, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Hu Y, Liu H, Zheng C, Li P, Xie J, Liu F, Li Z, Zhao G, Yang K, Liu C, Li H, Chen P, Ji J, Li G; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Effect of Laparoscopic vs Open Distal Gastrectomy on 3-Year Disease-Free Survival in Patients With Locally Advanced Gastric Cancer: The CLASS-01 Randomized Clinical Trial. JAMA. 2019 May 28;321(20):1983-1992. doi: 10.1001/jama.2019.5359. PMID 31135850
- [Background] Deng ZJ, Nie RC, Lu J, Chen XJ, Xiang J, Huang CM, Chen YB, Peng JS, Chen S. Survival analysis of stage II gastric cancer patients after D2 gastrectomy: a Chinese people-based research. BMC Gastroenterol. 2021 Oct 7;21(1):363. doi: 10.1186/s12876-021-01937-9. PMID 34620108
- [Background] Li Q, Zhang X, Tang M, Song M, Zhang Q, Zhang K, Ruan G, Zhang X, Ge Y, Yang M, Liu Y, Xu H, Song C, Wang Z, Shi H. Different muscle mass indices of the Global Leadership Initiative on Malnutrition in diagnosing malnutrition and predicting survival of patients with gastric cancer. Nutrition. 2021 Sep;89:111286. doi: 10.1016/j.nut.2021.111286. Epub 2021 Apr 24. PMID 34090215
- [Background] Davis JL, Selby LV, Chou JF, Schattner M, Ilson DH, Capanu M, Brennan MF, Coit DG, Strong VE. Patterns and Predictors of Weight Loss After Gastrectomy for Cancer. Ann Surg Oncol. 2016 May;23(5):1639-45. doi: 10.1245/s10434-015-5065-3. Epub 2016 Jan 5. PMID 26732274
- [Background] Takahashi S, Shimizu S, Nagai S, Watanabe H, Nishitani Y, Kurisu Y. Characteristics of sarcopenia after distal gastrectomy in elderly patients. PLoS One. 2019 Sep 11;14(9):e0222412. doi: 10.1371/journal.pone.0222412. eCollection 2019. PMID 31509590
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Kawamura T, Makuuchi R, Tokunaga M, Tanizawa Y, Bando E, Yasui H, Aoyama T, Inano T, Terashima M. Long-Term Outcomes of Gastric Cancer Patients with Preoperative Sarcopenia. Ann Surg Oncol. 2018 Jun;25(6):1625-1632. doi: 10.1245/s10434-018-6452-3. Epub 2018 Apr 9. PMID 29633095
- [Background] Lee JK, Park YS, Lee K, Youn SI, Won Y, Min SH, Ahn SH, Park DJ, Kim HH. Prognostic significance of surgery-induced sarcopenia in the survival of gastric cancer patients: a sex-specific analysis. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1897-1907. doi: 10.1002/jcsm.12793. Epub 2021 Sep 17. PMID 34533290
- [Background] Kudou K, Saeki H, Nakashima Y, Sasaki S, Jogo T, Hirose K, Hu Q, Tsuda Y, Kimura K, Nakanishi R, Kubo N, Ando K, Oki E, Ikeda T, Maehara Y. Postoperative development of sarcopenia is a strong predictor of a poor prognosis in patients with adenocarcinoma of the esophagogastric junction and upper gastric cancer. Am J Surg. 2019 Apr;217(4):757-763. doi: 10.1016/j.amjsurg.2018.07.003. Epub 2018 Jul 10. PMID 30005807
- [Background] Kudou K, Saeki H, Nakashima Y, Kimura K, Ando K, Oki E, Ikeda T, Maehara Y. Postoperative Skeletal Muscle Loss Predicts Poor Prognosis of Adenocarcinoma of Upper Stomach and Esophagogastric Junction. World J Surg. 2019 Apr;43(4):1068-1075. doi: 10.1007/s00268-018-4873-6. PMID 30478682
- [Background] Miyazaki Y, Omori T, Fujitani K, Fujita J, Kawabata R, Imamura H, Okada K, Moon JH, Hirao M, Matsuyama J, Saito T, Takahashi T, Kurokawa Y, Yamasaki M, Takiguchi S, Mori M, Doki Y; Osaka University Clinical Research Group for Gastroenterological Study. Oral nutritional supplements versus a regular diet alone for body weight loss after gastrectomy: a phase 3, multicenter, open-label randomized controlled trial. Gastric Cancer. 2021 Sep;24(5):1150-1159. doi: 10.1007/s10120-021-01188-3. Epub 2021 Apr 9. PMID 33835329
- [Background] Meng Q, Tan S, Jiang Y, Han J, Xi Q, Zhuang Q, Wu G. Post-discharge oral nutritional supplements with dietary advice in patients at nutritional risk after surgery for gastric cancer: A randomized clinical trial. Clin Nutr. 2021 Jan;40(1):40-46. doi: 10.1016/j.clnu.2020.04.043. Epub 2020 Jun 2. PMID 32563598